CLINICAL TRIAL: NCT00270634
Title: A Phase IIb, Randomized, Multicenter, Open-Label, Concentration Controlled, Safety Study of ISA247 (Voclosporin) and Tacrolimus (Prograf®) in De Novo Renal Transplant Patients
Brief Title: Study of ISA247 (Voclosporin) in De Novo Renal Transplantation
Acronym: PROMISE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISA05-01
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Diseases
Keywords: Randomized Controlled Trials; Immunosuppression; Adult; Kidney Transplantation; Treatment Outcome
MeSH Terms: conditions — Kidney Diseases | interventions — voclosporin; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Dose Voclosporin (Active Comparator): Low dose voclosporin
  Interventions: Drug: Voclosporin
- Mid Dose Voclosporin (Active Comparator): Mid Dose Voclosporin
  Interventions: Drug: Voclosporin
- High Dose Voclosporin (Active Comparator): High Dose Voclosporin
  Interventions: Drug: Voclosporin
- Tacrolimus (Active Comparator): Standard Dose Tacrolimus
  Interventions: Drug: tacrolimus

INTERVENTIONS:
Drug: Voclosporin — voclosporin 0.4, 0.6, 0.8 mg/kg po BID
  Other Names: ISA247
  Arms: High Dose Voclosporin; Low Dose Voclosporin; Mid Dose Voclosporin
Drug: tacrolimus — tacrolimus 0.05 mg/kg po BID
  Arms: Tacrolimus

SUMMARY:
This study will see if voclosporin is safe and effective in preventing kidney transplant rejection.

DETAILED DESCRIPTION:
Prograf® (tacrolimus) is associated with numerous side effects, including neurotoxicity, nephrotoxicity, polyoma nephropathy, QT prolongation, and New Onset Diabetes Mellitus After Transplant (NODAT). Voclosporin is a novel calcineurin inhibitor intended for use in the prevention of organ graft rejection.

Comparison(s): Voclosporin at 3 dose levels (0.4, 0.6, and 0.8 mg/kg twice a day) compared to tacrolimus

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 - 65 years inclusive at the time of screening.
* Patients must be receiving a first cadaveric or living donor renal transplant.
* Patients must be able to receive oral medication at time of randomization.
* Females who are not pregnant or nursing or planning to become pregnant during the course of the study, or 3 months after last dose of study medication.
* Sexually-active women of child-bearing potential (including those who are < 1 year postmenopausal) and sexually-active men who are practicing a highly effective method of birth control. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly and will include implants, injectables, combined oral contraceptives, double-barrier method, sexual abstinence, or a sterile partner. Sexually-active men and women of child-bearing potential should continue to practice contraception as outlined above during treatment and for ≥ 3 months after the last dose of voclosporin.
* Able to give written informed consent prior to screening procedures.
* Able to keep study appointments and cooperate with all study requirements, in the opinion of the investigator.

Exclusion Criteria:

* Receiving a HLA (human leukocyte antigen)identical living related transplant.
* Cold ischemic time > 24 hours.
* Peak PRA (panel reactive antibodies) > 30%
* Cadaveric donors who are over age 60, non-heart beating donors, or any cadaveric donors positive for HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV).
* Transplantation of multiple grafts (e.g. kidney and pancreas).
* Systemic infections requiring continued therapy at the time of entry into this study. (Prophylaxis against cytomegalovirus [CMV] and/or pneumocystis carinii pneumonia (PCP) infection will be permitted).
* Serologic evidence or known latent human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C (HCV) virus. Known negative serology prior to study entry may be used.
* A current malignancy or history of malignancy within 5 years or a history of lymphoma at any time. Subjects can be enrolled with a history of squamous or basal cell carcinoma that has been surgically excised or removed with curettage and electrodesiccation.
* Requires prohibited medications or treatment during the study.
* Alanine transaminase (ALT), aspartate transaminase (AST), or gamma-glutamyl transferase (GGT) ≥ 3x upper limit of normal (ULN) at time of transplantation.
* White blood cell count ≤ 2.8 x 10^9/L.
* Triglycerides ≥ 3x ULN.
* Pregnant women or nursing mothers.
* Has used any investigational drug or device within 28 days or 5 half lives (whichever is longer) prior to enrollment.
* Previous exposure to voclosporin.
* A history of active alcoholism or drug addiction within 1 year prior to study entry.
* Weighs < 45 kg (99 lbs) or > 140 kg (308 lbs).
* A history of disease, including mental/emotional disorder that would interfere with the subject's participation in the study, or that might cause the administration of voclosporin to pose a significant risk to the subject, in the opinion of the investigator.
* Allergy to iodine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2006-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Abramowicz, MD, PhD, Study Director — Erasme University Hospital; Philip Belitsky, MD, Study Director — No Affiliation; Arthur Matas, MD, Study Director — University of Minnesota; Mark Pescovitz, MD, Study Director — Indiana University; A. Osama Gaber, MD, Study Director — The Methodist Hospital Research Institute
Locations (37):
- United States (32):
  - Isotechnika Investigational Site, Birmingham, Alabama
  - Isotechnika Investigational Site, Los Angeles, California
  - Isotechnika Investigational Site, Orange, California
  - Isotechnika Investigational Site, Palo Alto, California
  - Isotechnika Investigational Site, San Diego, California
  - Isotechnika Investigational Site, San Francisco, California
  - Isotechnika Investigational Site, Denver, Colorado
  - Isotechnika Investigational Site, Gainesville, Florida
  - Isotechnika Investigational Site, Tampa, Florida
  - Isotechnika Investigational Site, Chicago, Illinois
  - Isotechnika Investigational Site, Lexington, Kentucky
  - Isotechnika Investigational Site, New Orleans, Louisiana
  - Isotechnika Investigational Site, Baltimore, Maryland
  - Isotechnika Investigational Site, Boston, Massachusetts
  - Isotechnika Investigational Site, Ann Arbor, Michigan
  - Isotechnika Investigational Site, Detroit, Michigan
  - Isotechnika Investigational Site, Rochester, Minnesota
  - Isotechnika Investigational Site, Livingston, New Jersey
  - Isotechnika Investigational Site, Buffalo, New York
  - Isotechnika Investigational Site, Hawthorne, New York
  - Isotechnika Investigational Site, New York, New York
  - Isotechnika Investigational Site, Rochester, New York
  - Isotechnika Investigational Site, Durham, North Carolina
  - Isotechnika Investigational Site, Winston-Salem, North Carolina
  - Isotechnika Investigational Site, Cincinnati, Ohio
  - Isotechnika Investigational Site, Portland, Oregon
  - Isotechnika Investigational Site, Philadelphia, Pennsylvania
  - Isotechnika Investigational Site, Charleston, South Carolina
  - Isotechnika Investigational Site, Memphis, Tennessee
  - Isotechnika Investigational Site, Dallas, Texas
  - Isotechnika Investigational Site, Houston, Texas
  - Isotechnika Investigational Site, Richmond, Virginia
- Canada (5):
  - Isotechnika Investigational Site, Edmonton, Alberta
  - Isotechnika Investigational Site, London, Ontario
  - Isotechnika Investigational Site, Toronto, Ontario
  - Isotechnika Investigational Site, Montreal, Quebec
  - Isotechnika Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Gregory CR, Kyles AE, Bernsteen L, Wagner GS, Tarantal AF, Christe KL, Brignolo L, Spinner A, Griffey SM, Paniagua RT, Hubble RW, Borie DC, Morris RE. Compared with cyclosporine, ISATX247 significantly prolongs renal-allograft survival in a nonhuman primate model. Transplantation. 2004 Sep 15;78(5):681-5. doi: 10.1097/01.tp.0000131950.75697.71. PMID 15371668
- [Background] Stalder M, Birsan T, Hubble RW, Paniagua RT, Morris RE. In vivo evaluation of the novel calcineurin inhibitor ISATX247 in non-human primates. J Heart Lung Transplant. 2003 Dec;22(12):1343-52. doi: 10.1016/s1053-2498(03)00033-0. PMID 14672749
- [Background] Abel MD, Aspeslet LJ, Freitag DG, Naicker S, Trepanier DJ, Kneteman NM, Foster RT, Yatscoff RW. ISATX247: a novel calcineurin inhibitor. J Heart Lung Transplant. 2001 Feb;20(2):161. doi: 10.1016/s1053-2498(00)00290-4. No abstract available. PMID 11250240
- [Result] Busque S, Cantarovich M, Mulgaonkar S, Gaston R, Gaber AO, Mayo PR, Ling S, Huizinga RB, Meier-Kriesche HU; PROMISE Investigators. The PROMISE study: a phase 2b multicenter study of voclosporin (ISA247) versus tacrolimus in de novo kidney transplantation. Am J Transplant. 2011 Dec;11(12):2675-84. doi: 10.1111/j.1600-6143.2011.03763.x. Epub 2011 Sep 22. PMID 21943027
- [Derived] Mayo PR, Ling SY, Huizinga RB, Freitag DG, Aspeslet LJ, Foster RT. Population PKPD of voclosporin in renal allograft patients. J Clin Pharmacol. 2014 May;54(5):537-45. doi: 10.1002/jcph.237. Epub 2013 Nov 30. PMID 24243422

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 334 de novo renal transplant patients were recruited in 36 US and 4 Canadian transplant centres between January 2006 and December 2007.
Pre-assignment Details: PROMISE was open to adult recipients of a first deceased or living donor renal transplant. Patients with established renal function (as demonstrated by urine output of at least 40 mL/h and a decline of creatinine of at least 15% from baseline during the first 24 h post-transplant) were randomized.
Groups:
- High Dose Voclosporin: High Dose Voclosporin: Initial dose of 0.8 mg/kg po BID
- Mid Dose Voclosporin: Mid Dose Voclosporin: Initial dose of 0.6 mg/kg po BID
- Low Dose Voclosporin: Low dose voclosporin: Initial dose of 0.4 mg/kg po BID
- Tacrolimus: Standard Dose Tacrolimus: Initial dose of 0.05 mg/kg po BID
Period: Overall Study
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Started | 87 | 77 | 84 | 86
Completed | 70 | 64 | 62 | 81
Not Completed | 17 | 13 | 22 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus | Total
Number analyzed (Participants) | 87 | 77 | 84 | 86 | 334
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 82 | 76 | 79 | 82 | 319
  >=65 years | 5 | 1 | 5 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 33 | 31 | 113
  Male | 63 | 52 | 51 | 55 | 221
Region of Enrollment [Number; unit: participants]
  United States | 74 | 67 | 74 | 75 | 290
  Canada | 13 | 10 | 10 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: Biopsy Proven Acute Rejection (BPAR)
Description: The primary objective of the PROMISE trial was to demonstrate noninferiority of biopsy proven acute rejection (BPAR) rate in de novo renal transplant patients at 6 months in at least one VCS treatment group.
Time Frame: Six months
Measure: Number; unit: percentage of participants
Groups:
- High Dose Voclosporin: Starting dose of 0.8 mg/kg
- Mid Dose Voclosporin: Starting dose of 0.6 mg/kg
- Low Dose Voclosporin: Starting dose of 0.4 mg/kg
- Tacrolimus: Standard dose
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Number analyzed (Participants) | 87 | 77 | 84 | 86
percentage of participants | 2.3 [upper limit 1.3] | 9.1 [upper limit 10.8] | 10.7 [upper limit 11.4] | 5.8 [0 to 0]
Statistical Analysis 1: Comparison: High Dose Voclosporin vs Tacrolimus; The 6-month BPAR rate was used to calculate an estimate of the difference in rates between each VCS group and TAC, combining across pooled investigative center strata, weighted by the number of patients in each of the pooled center strata. The overall standard error was estimated for the linear combination of proportions. Using this statistic and its standard error, the upper bound one-sided 95% C.I. was constructed for the difference in BPAR rates between groups (VCS - TAC); Test type: Non-Inferiority or Equivalence — The sample size was determined holding the probability of a type-I error at a = 0.05, and the power at 0.76. The rate of BPAR at 6 months posttransplant was assumed to be 0.20 in the control arm, and the noninferiority margin was chosen to be -0.15. A sample size for this phase-2b trial is determined to be 76 subjects in each dose group or a total of 304 patients. Assuming a 10% dropout rate during the study, ∼332 subjects were to be proportionally randomized in this study; t-test, 1 sided; Weighted Average Difference = -3.2, 95% CI 1-sided [upper limit 1.3] — The upper bound of the confidence interval was a measure of non-inferiority of VCS to TAC. VCS was considered non-inferior to TAC if the upper one-sided 95% confidence bound was less than 15%
Statistical Analysis 2: Comparison: Mid Dose Voclosporin vs Tacrolimus; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; t-test, 1 sided; Weighted Average Difference = 4.6, 95% CI 1-sided [upper limit 10.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Low Dose Voclosporin vs Tacrolimus; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; t-test, 1 sided; Weighted Average Difference = 4.9, 95% CI 1-sided [upper limit 11.4] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: To Demonstrate a 5% Improvement in Renal Function as Measured by Iothalamate Glomerular Filtration Rate (GFR)
Description: ANOVAs to test for differences in GFR at Month 6.
Time Frame: Six months
Population: Standard deviation around Iothalamate GFR made results uninterpretable, therefore Nankivell GFR was reported as it was collected a priori.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Number analyzed (Participants) | 87 | 77 | 84 | 86
mL/min | 68 (13) | 72 (12) | 71 (13) | 69 (29)

3. Secondary Outcome: The Pharmacokinetic-pharmacodynamic Relationship Between Voclosporin and Calcineurin Inhibition (CNi), or Tacrolimus and Calcineurin Inhibition
Description: A sparse sampling protocol of whole blood samples obtained on Day 180 at time points immediately prior to drug administration and at 1, 2, and 4 hours post-dose were utilized.
  Standard non-compartmental analysis (NCA) was performed on whole blood concentration data for voclosporin and its metabolites, tacrolimus, MPA (mycophenolic acid) and MPAG (mycophenolic acid glucuronide). Tmax and Cmax were obtained directly from the concentration-time profiles without interpolation. AUC(0-4)[area under the curve] was calculated using log-linear trapezoidal rule. Cmax, AUC(0-4), C0 and C2 were summarized using descriptive statistics.
Time Frame: Six months
Population: For subjects participating in the PK/PD portion of the study, a calcineurin sample was drawn prior to drug administration in order to assess baseline calcineurin levels. Blood samples were taken at Month 6 for the assessment of pharmacokinetics and pharmacodynamics. Participation by subjects was optional.
Measure: Mean (Standard Deviation); unit: % Calcineurin (CNi) compared to baseline
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Number analyzed (Participants) | 33 | 25 | 20 | 28
% Calcineurin (CNi) compared to baseline | 57.3 (14.4) | 47.5 (16.4) | 38.8 (16.3) | 23.0 (13.8)

4. Secondary Outcome: Patient Survival
Time Frame: Six months
Measure: Number; unit: Percentage of patients
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Number analyzed (Participants) | 87 | 77 | 84 | 86
Percentage of patients | 98.9 | 100 | 100 | 97.7

5. Secondary Outcome: Graft Survival
Time Frame: Six months
Measure: Number; unit: Percentage of patients
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Number analyzed (Participants) | 87 | 77 | 84 | 86
Percentage of patients | 98.9 | 100 | 100 | 97.7

6. Secondary Outcome: Hypertension, Hyperlipidemia, or Hyperglycemia
Time Frame: Six months
Population: Endpoint
Measure: Number; unit: Percentage of patients
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Number analyzed (Participants) | 87 | 77 | 84 | 86
Percentage of patients
  Treatment with an Antihypertensive | 96.6 (1) | 97.4 (1) | 96.4 (1.2) | 95.3 (1.2)
  Triglyceride values > ULN | 28 (18) | 30 (18) | 18 (22) | 39 (16)
  New Onset of Diabetes Mellitus After Transplant | 17.7 | 5.7 | 1.6 | 16.4

7. Secondary Outcome: A Composite of Biopsy-proven Chronic Rejection Graft Loss, Death, or Lost to Follow up.
Time Frame: Six months
Population: Per Protocol Dataset
Measure: Number; unit: Percentage of patients
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Number analyzed (Participants) | 54 | 54 | 54 | 76
Percentage of patients | 5.6 | 7.4 | 3.7 | 3.9

ADVERSE EVENTS:
Time Frame: 6 month treatment
Description: AEs were assessed at each clinic visit throughout the study.
Arm/Group | High Dose Voclosporin | Mid Dose Voclosporin | Low Dose Voclosporin | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 40/87 | 35/77 | 36/84 | 37/86
Other Adverse Events (participants affected / at risk) | 84/87 | 76/77 | 83/84 | 85/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Voclosporin (N=87) | Mid Dose Voclosporin (N=77) | Low Dose Voclosporin (N=84) | Tacrolimus (N=86)
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphocele (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 0 | 1
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Unstable Angina (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Strangulated Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarhhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal Ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peridontal Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 0 | 3
Kidney Transplant Rejection (Immune system disorders) | 4 | 10 | 18 | 6
Transplant Rejection (Immune system disorders) | 0 | 0 | 1 | 0
Abcess Limb (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridial Infection (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus Infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterococcal Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Gastritis Viral (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 2
Hepatitis A (Infections and infestations) | 0 | 0 | 1 | 0
Localized Infection (Infections and infestations) | 1 | 0 | 0 | 0
Oesophageal Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Polyomavirus-Associated Nephropathy (Infections and infestations) | 0 | 1 | 1 | 0
Post Operative Wound Infection (Infections and infestations) | 0 | 1 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 0 | 1
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Complications of Transplanted Kidney (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Perinephric Collection (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Renal Haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Renal Lymphocele (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Urinary Anastomotic Leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post Procedural Urine Leak (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 6 | 3 | 3 | 3
Electrocardiogram ST Segment Abnormal (Investigations) | 1 | 0 | 0 | 0
International Normalised Ratio Decreased (Investigations) | 0 | 0 | 0 | 2
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0 | 3
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Papillary Tumour of Renal Pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Anoxic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Neurological Symptom (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Acute Psychotic (Psychiatric disorders) | 0 | 0 | 0 | 1
Paranoia (Psychiatric disorders) | 0 | 1 | 0 | 0
Anastomotic Stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Complications of Transplanted Kidney (Renal and urinary disorders) | 1 | 0 | 0 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 4 | 0 | 2
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal Vein Thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urethral Obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Benign Prostatic Hyperplagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cyst Drainage (Surgical and medical procedures) | 1 | 0 | 0 | 0
Lymphocele Marsupialisation (Surgical and medical procedures) | 0 | 1 | 1 | 0
Nephrectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
Steal Syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Subclavian Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose Voclosporin (N=87) | Mid Dose Voclosporin (N=77) | Low Dose Voclosporin (N=84) | Tacrolimus (N=86)
ANAEMIA (Blood and lymphatic system disorders) | 27 | 24 | 30 | 27
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 7 | 4 | 2 | 4
LEUKOPENIA (Blood and lymphatic system disorders) | 13 | 15 | 14 | 12
TACHYCARDIA (Cardiac disorders) | 6 | 4 | 9 | 7
EAR PAIN (Ear and labyrinth disorders) | 0 | 0 | 0 | 6
HYPERCALCAEMIA (Endocrine disorders) | 5 | 7 | 4 | 3
VISION BLURRED (Eye disorders) | 5 | 4 | 1 | 3
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 | 5 | 13 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 12 | 9 | 8 | 7
CONSTIPATION (Gastrointestinal disorders) | 35 | 34 | 43 | 31
DIARRHOEA (Gastrointestinal disorders) | 31 | 29 | 16 | 43
DYSPEPSIA (Gastrointestinal disorders) | 10 | 6 | 8 | 18
FLATULENCE (Gastrointestinal disorders) | 6 | 2 | 3 | 5
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 | 4 | 6 | 5
NAUSEA (Gastrointestinal disorders) | 36 | 28 | 36 | 35
VOMITING (Gastrointestinal disorders) | 14 | 14 | 13 | 19
ASTHENIA (General disorders) | 4 | 2 | 4 | 8
CHEST PAIN (General disorders) | 8 | 4 | 3 | 8
CHILLS (General disorders) | 4 | 1 | 5 | 5
FATIGUE (General disorders) | 16 | 11 | 21 | 12
OEDEMA (General disorders) | 20 | 21 | 20 | 15
OEDEMA PERIPHERAL (General disorders) | 28 | 31 | 24 | 23
PAIN (General disorders) | 6 | 7 | 3 | 1
PYREXIA (General disorders) | 15 | 9 | 10 | 13
KIDNEY TRANSPLANT REJECTION (Immune system disorders) | 4 | 4 | 7 | 2
CANDIDIASIS (Infections and infestations) | 5 | 3 | 3 | 3
NASOPHARYNGITIS (Infections and infestations) | 6 | 5 | 2 | 2
SINUSITIS (Infections and infestations) | 6 | 4 | 1 | 3
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 3 | 7 | 5
URINARY TRACT INFECTION (Infections and infestations) | 11 | 4 | 5 | 6
INCISION SITE COMPLICATION (Injury, poisoning and procedural complications) | 17 | 20 | 25 | 22
PERINEPHRIC COLLECTION (Injury, poisoning and procedural complications) | 6 | 2 | 4 | 3
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 29 | 28 | 28 | 30
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 5
BLOOD CREATININE INCREASED (Investigations) | 20 | 11 | 20 | 10
BLOOD PRESSURE INCREASED (Investigations) | 5 | 3 | 2 | 3
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 4 | 5 | 5
URINE OUTPUT DECREASED (Investigations) | 5 | 1 | 3 | 4
WEIGHT INCREASED (Investigations) | 10 | 12 | 11 | 12
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 3 | 1 | 5
GOUT (Metabolism and nutrition disorders) | 2 | 5 | 0 | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 5 | 3 | 2 | 7
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 15 | 16 | 14 | 20
HYPERKALAEMIA (Metabolism and nutrition disorders) | 25 | 17 | 12 | 22
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 6 | 14 | 9 | 9
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 | 3 | 5 | 7
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 10 | 3 | 8 | 10
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14 | 9 | 12 | 13
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 34 | 21 | 22 | 37
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 28 | 32 | 32 | 34
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 4 | 6 | 4 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 9 | 13 | 9
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 11 | 6 | 5 | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 5
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7 | 8 | 6 | 7
DIZZINESS (Nervous system disorders) | 9 | 8 | 13 | 12
HEADACHE (Nervous system disorders) | 14 | 12 | 16 | 12
PARAESTHESIA (Nervous system disorders) | 5 | 7 | 6 | 6
TREMOR (Nervous system disorders) | 18 | 22 | 10 | 24
ANXIETY (Psychiatric disorders) | 7 | 6 | 9 | 7
INSOMNIA (Psychiatric disorders) | 20 | 20 | 19 | 33
DYSURIA (Renal and urinary disorders) | 11 | 5 | 8 | 8
HAEMATURIA (Renal and urinary disorders) | 8 | 11 | 14 | 6
HYDRONEPHROSIS (Renal and urinary disorders) | 4 | 4 | 1 | 6
PROTEINURIA (Renal and urinary disorders) | 4 | 2 | 5 | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 11 | 7
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14 | 9 | 12 | 17
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 2 | 2
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 4 | 6
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 3 | 2
ACNE (Skin and subcutaneous tissue disorders) | 2 | 4 | 6 | 4
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 5 | 2 | 7
HAIR GROWTH ABNORMAL (Skin and subcutaneous tissue disorders) | 3 | 6 | 6 | 0
HYPERTRICHOSIS (Skin and subcutaneous tissue disorders) | 5 | 5 | 2 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 7 | 6 | 6 | 13
RASH (Skin and subcutaneous tissue disorders) | 8 | 9 | 7 | 8
INCISIONAL DRAINAGE (Surgical and medical procedures) | 3 | 1 | 5 | 1
WOUND DRAINAGE (Surgical and medical procedures) | 2 | 4 | 3 | 5
HYPERTENSION (Vascular disorders) | 23 | 23 | 29 | 26
HYPOTENSION (Vascular disorders) | 8 | 4 | 9 | 12

LIMITATIONS AND CAVEATS:
By limiting access to patients at relatively low risk for rejection and no delayed graft function, the results observed may not be applicable to all renal transplant recipients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days